CLINICAL TRIAL: NCT03552003
Title: Prospective Study on Elderly (≥ 65 Years) Patients Affected With Classical Hodgkin Lymphoma Undergoing Comprehensive Geriatric Assessment at Diagnosis
Brief Title: Study for Elderly (≥ 65 Years) Patients With Classical Hodgkin Lymphoma Undergoing CGA at Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_ELDHL
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: Hodgkin; Elderly patients; CGA
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mandatory:
  1) paraffin block for diagnosis review
  Optional:
  1. paraffin block for TISSUE MICRO ARRAYS analyses
  2. 3ml blood adsorbed on a swab tip for IMMUNO SENESCENCE AND FRAILTY evaluation
  3. 3ml blood adsorbed on a swab tip for IMMUNO SENESCENCE AND TORQUE TENO VIRUS evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly diagnosed elderly cHL patients: Newly diagnosed elderly cHL patients undergoing CGA before any therapy (treatment for clinical practise) with the use of ADL, IADL and CIRS-G. Patients who will be considered not eligible to receive treatment or to be given only palliative therapy after CGA assessment are eligible for the study
  Interventions: Other: Treatment for clinical practise

INTERVENTIONS:
Other: Treatment for clinical practise — Prospective data collection with the aim to to develop a prognostic index for elderly patients with newly diagnosed cHL

SUMMARY:
The aim of the study is to develop a prognostic index for elderly patients with newly diagnosed cHL starting from a prospective observational study of consecutive cases registered after the completion of the Comprehensive Geriatric Assessment (CGA)

DETAILED DESCRIPTION:
The aim of the study is to develop a prognostic index for elderly patients with newly diagnosed cHL starting from a prospective observational study of consecutive cases registered after the completion of the Comprehensive Geriatric Assessment (CGA) Prospective data collection study of a consecutive series of newly diagnosed elderly cHL patients undergoing CGA before any therapy with the use of ADL, IADL and CIRS-G. Patients who will be considered not eligible to receive treatment or to be given only palliative therapy after CGA assessment are eligible for the study. Patients will be screened and restaged according to clinical practice instrumental and laboratory assessments timing and type of examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of classical Hodgkin Lymphoma
2. Age ≥ 65 year
3. Evaluation of Comprehensive Geriatric Assessment at baseline
4. Signed informed consent
5. Previously untreated patients

Exclusion Criteria:

None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: newly diagnosed elderly cHL patients undergoing CGA before any therapy with the use of ADL, IADL and CIRS-G. Patients who will be considered not eligible to receive treatment or to be given only palliative therapy after CGA assessment are eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
OS | June 2018-December 2025 (7.5 years)
  Overall survival (OS). From the date of diagnosis to the date of last observation or death from any cause

SECONDARY OUTCOMES:
PFS | June 2018-December 2025 (7.5 years)
  Progression Free Survival (PFS): From the date of diagnosis to the last follow-up, or to one of the following events: disease progression during treatment, or relapse, or death from any cause.
FFS | June 2018-December 2025 (7.5 years)
  Failure Free Survival (FFS). From the date of diagnosis to to any treatment failure including disease progression, or discontinuation of treatment for any reason, (eg, disease progression, toxicity, patient preference, initiation of new treatment), or death from any cause.
Response initial therapy | June 2018-January 2024 (5.5 years, 6-7 month after the enrolment)
  Response initial therapy: Rate of complete remission (CR) after chemotherapy +/-RT, according to Cheson 2007

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Ruggero Zilioli, MD, Principal Investigator — SC Ematologia, ASST Grande Ospedale Metropolitano Niguarda, Milano - Italy
Locations (44):
- Italy (44):
  - SC Ematologia AO SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Università Politecnica delle Marche - Clinica di Ematologia, Ancona
  - Azienda Ospedaliera S. Giuseppe Moscati - S.C. Ematologia e Trapianto emopoietico, Avellino
  - Centro Riferimento Oncologico - S.O.C. Oncologia Medica A, Aviano
  - AOU Policlinico Consorziale - U.O. Ematologia con Trapianto, Bari
  - Ospedale "Monsignor Raffaele Dimiccoli" - Ematologia, Barletta
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Ospedale Businco - Ematologia, Cagliari
  - Università Cattolica del Sacro Cuore - Ematologia, Campobasso
  - Ospedale di Castelfranco Veneto - Ematologia, Castelfranco Veneto
  - Azienda Ospedaliera di Cosenza - UOC Ematologia, Cosenza
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - UOC Ematologia PO Spaziani, Frosinone
  - Ospedali Riuniti del Canavese - S.C. Medicina trasfusionale ed Ematologia, Ivrea
  - Ospedale Madonna delle Grazie - Ematologia, Matera
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) - Ematologia, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano - Ematologia, Milan
  - Istituto Scientifico San Raffaele - Unità Linfomi - Dipartimento Oncoematologia, Milan
  - Ospedale Maggiore Policlinico - Fondazione IRCCS Ca' Granda - Ematologia, Milan
  - AOU Università degli Studi della Campania Luigi Vanvitelli - Oncologia Medica ed Ematologia, Napoli
  - AOU Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - AOU di Padova - Ematologia, Padua
  - I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1, Padua
  - AOU Policlinico Giaccone - Ematologia, Palermo
  - AOU di Parma - UO Ematologia e CTMO, Parma
  - IRCCS Policlinico S. Matteo di Pavia - Div. di Ematologia, Pavia
  - Ospedale S. Maria della Misericordia - Ematologia, Perugia
  - Ospedale Guglielmo da Saliceto - U.O. Ematologia, Piacenza
  - Ospedale delle Croci - Ematologia, Ravenna
  - Azienda Unità Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia, Reggio Emilia
  - Ospedale degli Infermi di Rimini - U.O. di Ematologia, Rimini
  - AO Sant'Andrea - Ematologia, Roma
  - Ospedale S. Camillo - Ematologia, Roma
  - Università Cattolica S. Cuore - Ematologia, Roma
  - Istituto Clinico Humanitas - U.O. Ematologia, Rozzano
  - Nuovo Ospedale Civile di Sassuolo - Day Hospital Oncologico, Sassuolo
  - AOU Senese - U.O.C. Ematologia, Siena
  - Azienda Ospedaliera della Valtellina e della Valchiavenna P.O. Sondrio - Medicina Interna - Centro Malattie del Sangue P.O. Sondrio, Sondrio
  - A.O. S. Maria di Terni - S.C. Oncoematologia, Terni
  - A.O.U. Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - A.O.U. Citta della Salute e della Scienza di Torino - S.C. Ematologia, Torino
  - Ospedale Ca Foncello - S.C di Ematologia, Treviso
  - A.O. C. Panico - U.O.C Ematologia e Trapianto, Tricase